CLINICAL TRIAL: NCT06878937
Title: 'Thriving With Bipolar Disorder': Co-design and Pilot Evaluation of a Peer-Delivered, Quality of Life Focused Group Psychoeducation Program
Brief Title: 'Thriving With Bipolar Disorder': Co-design and Evaluation of a Peer-Led Education Program Focused on Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mood Disorders Association of Ontario (Unknown)
Responsible Party: Principal Investigator, Erin Michalak, Professor, Department of Psychiatry, Faculty of Medicine, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-03489
Record Dates: First submitted 2025-03-04; First posted 2025-03-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder (BD); Quality of Life (QOL)
Keywords: Psychoeducation; Peer-Support; Bipolar Disorder; Quality of Life; Self-Management
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Evaluation of the psychoeducation program will be conducted as a single-arm, uncontrolled, pilot feasibility trial. An explanatory sequential mixed-methods design will be used (Creswell & Clark, 2011).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer-Delivered Psychoeducation Program (Experimental): Individuals in this arm will complete the peer-delivered psychoeducation program.
  Interventions: Behavioral: Peer Delivered Psychoeducation Program

INTERVENTIONS:
Behavioral: Peer Delivered Psychoeducation Program — The peer delivered psychoeducation program is the only intervention being tested in this pilot evaluation study.

SUMMARY:
Self-management strategies can be used by individuals with bipolar disorder (BD) to cope with symptoms and improve quality of life (QoL). Peer-facilitated education programs have the potential to diversify delivery of self-management information by capitalizing on the expertise of individuals who live well with BD. We have co-designed a novel, peer-facilitated, QoL-focused, group education program for people living with BD. This project will involve administration of the program and an evaluation of the feasibility, acceptability, and efficacy of this program for self-management of BD.

DETAILED DESCRIPTION:
Background and Purpose:

Peer support (where individuals with shared lived experience of a mental health condition provide each other with informational, emotional, and social support) may be an acceptable way to disseminate information on self-management strategies, capitalizing on the expertise and knowledge of people who live well with BD.

Peer-facilitated group psychoeducation includes the benefits of evidence-based self-management information and tools, with the added advantage of providing role models for recovery and modelling of self-management skills. Unfortunately, there is a dearth of BD-specific peer-facilitated self-management psychoeducation programs, and corresponding evaluations of their efficacy.

To capitalize on the potential of peer support to enhance the delivery of BD self-management information, content from two, web-based, self-directed psychoeducational interventions was adapted to create a peer-facilitated psychoeducation program using a community-based participatory research (CBPR) framework. The resulting program contains eight, weekly, two-hour sessions. Each session focuses on a topic related to QoL in BD (including Mood, Sleep, Physical Health, Relationships, Money, Self-esteem, and Independence), and contains a combination of education, opportunities for peer-to-peer knowledge exchange, and activities that facilitate practice of self-management strategies. A facilitator and attendee manual have been created for use in this program.

Methods:

The project will be implemented across two phases:

In the first phase, which we have already completed, we have applied CBPR principles to develop a peer-facilitated, QoL-focused group psychoeducation program for individuals with BD. The resulting program, entitled 'Thriving with bipolar disorder' will be delivered in eight, weekly, two-hour sessions that will be co-facilitated by two peer facilitators with lived experience of BD.

In the second phase, we will conduct a pilot evaluation of the feasibility, acceptability, and preliminary efficacy of the program. The program will be delivered through Hope+Me, an Ontario-based charity that supports people living with mood and anxiety disorders through education, advocacy, training, and support services. Four peer facilitators will be recruited through Hope+Me and will attend a ~5.5 hour training session prior to commencing the program. We will aim to recruit 32-40 program participants (8-10 per group) given previous research summarizing the ideal group size.

The evaluation will be conducted as a single-arm, uncontrolled, pilot feasibility trial. An explanatory sequential mixed-methods design will be used. The following data will be collected:

* Participants will provide baseline demographic and clinical information in a survey as part of their consent.
* Participants will complete surveys for efficacy measures at baseline, immediately after completing the program and 1 month after completing the program.
* Program feedback will be collected from participants immediately after completing the program through a Qualtrics survey.
* Peer facilitators will complete a brief, post-session Qualtrics survey each week, recording attendance, fidelity, and session feedback.

At the end of the intervention period, a subset of consenting participants (~n=12) and peer facilitators (~n=4) will be invited to participate in a one-hour qualitative individual interview over Zoom.

Study Population:

Four peer facilitators will be recruited through Hope+Me. We hope to recruit ~fourty program participants. Inclusion and exclusion criteria are specified in the 'Eligibility' section.

ELIGIBILITY:
Inclusion Criteria:

1. Program facilitators

   * aged 18 or older
   * a self-reported diagnosis of a mood disorder
   * sufficient access to an internet-enabled computer or smartphone device to access the Zoom teleconferencing platform
   * ability to understand, read and write English
   * at least one year of prior experience leading peer support groups or recovery programs through Hope+Me
   * previously received training through Hope+Me
   * completed a Criminal Records Check
2. Program participants

   * aged 18 or older
   * residing in Canada
   * a self-reported diagnosis of BD
   * ability to understand, read and write English
   * sufficient access to an internet-enabled computer or smartphone device to access the Zoom teleconferencing platform

Exclusion Criteria:

* inability to communicate in written and verbal English to a sufficient level to allow participation in the program and research activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Session Attendance) | Every week, from enrollment to the end of the intervention at 8 weeks.
  Feasibility will be assessed using program attendance rates. After each session, peer facilitators will complete a brief questionnaire to record the number of participants who attended each session. Feasibility is defined as the proportion of participants achieving the minimum attendance of 62.5% (i.e., five out of eight sessions), based on the median therapeutic dose in a review of group therapy program evaluations.

SECONDARY OUTCOMES:
Patient Health Questionnaire 8 (PHQ-8) | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Self-reported depressive symptoms will be assessed by the Patient Health Questionnaire-8 (PHQ-8), which evaluates 8 of the 9 criteria for depression from the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV). The eight Likert-type items ask about the frequency of depressive symptoms experienced in the past two weeks (0 = "Not at all" to 3 = "Nearly every day"). Responses are summed to create a total score (range: 0-24); higher scores indicate greater depression severity. The PHQ-8 performs comparably with clinician assessments; internal reliability has been demonstrated in population studies (Cronbach α=0.87).
  The PHQ-8 has comparable performance to the original nine item version (PHQ-9), which assesses all DSM-IV criteria, including current suicidal ideation. The PHQ-8 is chosen for this evaluation because this program doesn't incorporate formal psychiatric evaluation and supports, data collected is self-reported, and immediate follow-up isn't possible.
Quality of Life in Bipolar Disorder (QoL.BD) Scale | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  The Quality of Life in Bipolar Disorder (QoL.BD) Scale will be used to assess aspects of QoL specifically impacted by or relevant to BD. This scale assesses 12 core aspects of QoL (mood, sleep, physical health, cognition, household management, leisure, finances, relationships, self-esteem, spirituality, identity, and independence). Each domain contains four Likert-type items that assess satisfaction with that area (1 = Strongly Disagree to 5 = Strongly Agree). An overall score can be calculated by summing responses to the 48 items (range: 48-240), with higher scores indicating greater life satisfaction.
  During psychometric testing, the factor structure of the QoL.BD has been supported, and the scale has demonstrated excellent internal reliability (Cronbach α>0.8) and appropriate test-retest reliability. Construct validity has been supported through positive correlations with generic QoL instruments and negative correlations with depressive symptoms.
Altman Self-Rating Mania Scale | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Self-reported mania will be assessed using the Altman Self-Rating Mania Scale. This instrument measures behaviours and feelings during the past week using five items; a total score (range: 5-25) can be calculated by summing responses, with higher scores indicating more severe manic symptoms.
  Responses have been found to correlate strongly with clinician-rated mania; internal reliability is acceptable (Cronbach α>0.65).
Bipolar Recovery Questionnaire | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Personal recovery will be measured using the Bipolar Recovery Questionnaire. Items are informed by qualitative interviews regarding experiences of personal (as opposed to clinical) recovery in BD. This scale contains 36 visual analogue scales (range: 0-100); responses are summed to create an overall score (range: 0-3600). Higher scores are indicative of better self-appraised recovery.
  This instrument has been found to be internally consistent (Cronbach α=0.875) and reliable over a month-long test-retest period.
Stanford's Chronic Disease Self-Efficacy 'Manage Disease in General' Subscale | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Self-efficacy will be measured using the 5-item Manage Disease in General subscale of Stanford's Chronic Disease Self-Efficacy Scale. The score on this subscale is the mean of 5 Likert-type items (1 = not at all confident to 10 = totally confident). Higher scores on this subscale (range: 1-10) indicate greater confidence in managing the symptoms and impacts of a chronic health condition.
Self-Compassion Scale-Short Form | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Self-compassion will be measured using the Self-Compassion Scale-Short Form (61, 62), which contains 12 Likert-type items (1=Almost Never, 5 = Almost Always) used to assess 6 dimensions of self-compassion: self-kindness, self-judgement, common humanity, isolation, mindfulness, and overidentification. Subscales are calculated by averaging relevant items. To calculate an overall score (range: 1-5), negative subscales are reverse-coded. Higher overall scores indicate more frequent self-compassionate behaviours and attitudes.
  Internal consistency has been demonstrated (Cronbach α=0.86); confirmatory factor analysis supports both the 6 subscales and a single higher-order factor of self-compassion.
Internalised Stigma of Mental Illness Scale Brief Version | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Self-stigma will be measured using the Internalised Stigma of Mental Illness Scale Brief Version. This instrument contains 9 Likert-type items (1= Strongly Disagree, 4 = Strongly Agree); two are reverse-coded. Item responses are averaged for an overall score (range: 1-4); higher scores indicate more internalized stigmatizing attitudes towards mental illness.
  Internal consistency has been demonstrated (Cronbach α=0.86); confirmatory factor analysis supports a unidimensional factor structure.
Social Provisions Scale Short Form | At enrollment, immediately after the intervention at 8 weeks, and a follow-up 4 weeks after the intervention.
  Perceived social support will be measured using the Social Provisions Scale Short Form. This instrument contains 10 Likert-type items (1= Strongly Disagree, 4 = Strongly Agree) which evaluate an individual's perceptions of the availability of social support. An overall score (range: 10-40) and five subscales can be calculated by summing relevant items; subscales include guidance (receipt of information or advice), reliable alliance (practical help and support), reassurance of worth (feeling valued by others), attachment (emotional bonds), and social integration (sense of belonging to a group with shared interests and attitudes).
  Internal consistency of the scale has been supported (Cronbach α>0.80).
Client Satisfaction Questionnaire-8 | Immediately after the intervention at 8 weeks.
  The Client Satisfaction Questionnaire-8 will be used to assess attendees' satisfaction with the 'Thriving with Bipolar Disorder' program post-intervention.
  This instrument has high internal consistency (Cronbach α=0.91); higher scores have been associated with greater attendance of services and improved clinical outcomes
Group Climate Questionnaire Short Form | Every week, from enrollment to the end of the intervention at 8 weeks.
  To describe the acceptability of the group climate, we will use the Group Climate Questionnaire short form. This is the most widely used measure of group therapy cohesion, and can be completed by a group member, facilitator, or observer; here, to minimize response burden on attendees, weekly feedback will be provided by facilitators. It contains 12 items describing specific behaviours that are rated on a 7-point Likert scale (where 0 indicates "not at all" and 7 indicates "extremely"), three subscales can be calculated based on the mean score of relevant items. These subscales are Engaged (which describes a positive working group atmosphere), Avoiding (which describes avoidance of responsibility for group dynamics), and Conflict (which describes tension and anger between group members).
Feasibility (Fidelity) | Every week, from enrollment to the end of the intervention at 8 weeks.
  To evaluate fidelity, facilitators will self-report adherence to the manual using four self-report Likert-type items, asking them to report the degree to which they reviewed information as described in the manual, shared their own lived experiences, and facilitated group involvement in discussions and activities. This method of fidelity assessment was selected given that the use of external observers may impact participant willingness to participate in group discussions and activities. Similar self-reported fidelity assessments have previously been used in evaluations of peer-led programs.

OTHER OUTCOMES:
Program and Facilitator Feedback | Immediately after the intervention at 8 weeks.
  We will query attendee perceptions of program content, delivery, the facilitator, and the group environment, using a series of Likert-scale statements developed by the research team (1 = "Strongly Disagree" to 5 = "Strongly Agree"). Open-ended items will allow attendees to provide free-text feedback on program strengths and areas for improvement.
Qualitative Feedback | Immediately after the intervention at 8 weeks.
  Individual interviews (approximately one hour) will be conducted with a convenience sample of participants (~n=12) and facilitators (~n=4) post-intervention. A semi-structured interview guide will contain questions about the acceptability of program content and format, experiences of the group environment, perceptions of the facilitator, and changes experienced as a result of participation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any published articles after deidentification. Qualitative data will not be shared to protect privacy and confidentiality due to the potential risk of participant re-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after article publication.
Access Criteria: Researchers interested in using the data must provide a methodologically sound proposal. All requests should be directed to emma.morton@monash.edu. If a request is approved, the requesting party will need to secure behavioural research ethics board approval from their institution and sign a Clinical Study Data Transfer Agreement. Data will be shared using a secure file transfer service approved by the university (Microsoft OneDrive).
  The research team reserves the right to deny incomplete/inaccurate proposals, if there is a perceived conflict of interest, or if researchers cannot ensure sufficient measures are in place to maintain the security and privacy of the data.

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Biggs K, Hind D, Gossage-Worrall R, Sprange K, White D, Wright J, Chatters R, Berry K, Papaioannou D, Bradburn M, Walters SJ, Cooper C. Challenges in the design, planning and implementation of trials evaluating group interventions. Trials. 2020 Jan 29;21(1):116. doi: 10.1186/s13063-019-3807-4. PMID 31996259
- [Background] Tse S, Yuen WWY, Murray G, Davidson L, Lai Q, Kan A. Combining technical and expert-by-experience knowledge in the quest for personal recovery from bipolar disorder: a qualitative study. BMC Psychiatry. 2019 Nov 26;19(1):368. doi: 10.1186/s12888-019-2357-3. PMID 31771532
- [Background] Proudfoot J, Parker G, Manicavasagar V, Hadzi-Pavlovic D, Whitton A, Nicholas J, Smith M, Burckhardt R. Effects of adjunctive peer support on perceptions of illness control and understanding in an online psychoeducation program for bipolar disorder: a randomised controlled trial. J Affect Disord. 2012 Dec 15;142(1-3):98-105. doi: 10.1016/j.jad.2012.04.007. Epub 2012 Aug 2. PMID 22858215
- [Background] Shin C, Lee SH, Han KM, Yoon HK, Han C. Comparison of the Usefulness of the PHQ-8 and PHQ-9 for Screening for Major Depressive Disorder: Analysis of Psychiatric Outpatient Data. Psychiatry Investig. 2019 Apr;16(4):300-305. doi: 10.30773/pi.2019.02.01. Epub 2019 Apr 24. PMID 31042692
- [Background] Wu Y, Levis B, Riehm KE, Saadat N, Levis AW, Azar M, Rice DB, Boruff J, Cuijpers P, Gilbody S, Ioannidis JPA, Kloda LA, McMillan D, Patten SB, Shrier I, Ziegelstein RC, Akena DH, Arroll B, Ayalon L, Baradaran HR, Baron M, Bombardier CH, Butterworth P, Carter G, Chagas MH, Chan JCN, Cholera R, Conwell Y, de Man-van Ginkel JM, Fann JR, Fischer FH, Fung D, Gelaye B, Goodyear-Smith F, Greeno CG, Hall BJ, Harrison PA, Harter M, Hegerl U, Hides L, Hobfoll SE, Hudson M, Hyphantis T, Inagaki M, Jette N, Khamseh ME, Kiely KM, Kwan Y, Lamers F, Liu SI, Lotrakul M, Loureiro SR, Lowe B, McGuire A, Mohd-Sidik S, Munhoz TN, Muramatsu K, Osorio FL, Patel V, Pence BW, Persoons P, Picardi A, Reuter K, Rooney AG, Santos IS, Shaaban J, Sidebottom A, Simning A, Stafford L, Sung S, Tan PLL, Turner A, van Weert HC, White J, Whooley MA, Winkley K, Yamada M, Benedetti A, Thombs BD. Equivalency of the diagnostic accuracy of the PHQ-8 and PHQ-9: a systematic review and individual participant data meta-analysis. Psychol Med. 2020 Jun;50(8):1368-1380. doi: 10.1017/S0033291719001314. Epub 2019 Jul 12. PMID 31298180
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Morton E, Murray G, Yatham LN, Lam RW, Michalak EE. The Quality of Life in Bipolar Disorder (QoL.BD) questionnaire a decade on - A systematic review of the measurement of condition-specific aspects of quality of life in bipolar-disorder. J Affect Disord. 2021 Jan 1;278:33-45. doi: 10.1016/j.jad.2020.09.017. Epub 2020 Sep 7. PMID 32949871
- [Background] Morton E, Hou SH, Fogarty O, Murray G, Barnes S, Depp C; CREST.BD; Michalak E. A Web-Based Adaptation of the Quality of Life in Bipolar Disorder Questionnaire: Psychometric Evaluation Study. JMIR Ment Health. 2020 Apr 27;7(4):e17497. doi: 10.2196/17497. PMID 32338620
- [Background] Michalak EE, Murray G; Collaborative RESearch Team to Study Psychosocial Issues in Bipolar Disorder (CREST.BD). Development of the QoL.BD: a disorder-specific scale to assess quality of life in bipolar disorder. Bipolar Disord. 2010 Nov;12(7):727-40. doi: 10.1111/j.1399-5618.2010.00865.x. PMID 21040290
- [Background] MacKenzie, K. (1983). The clinical application of a group climate measure. In R.R. Dies & K.R. MacKenzie (Eds.), Advances in group psychotherapy: Integrating research and practice (pp. 159-170). International Universities Press.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Derived] Morton E, Kcomt A, Michalak EE. 'Thriving with bipolar disorder': The co-design of a peer-delivered group psychoeducation program and single-arm pilot feasibility evaluation protocol. PLoS One. 2025 Dec 17;20(12):e0338306. doi: 10.1371/journal.pone.0338306. eCollection 2025. PMID 41406148